CLINICAL TRIAL: NCT04120597
Title: Clinical and Basic Research on the Treatment of Zishen Qingre Lishi Huayu Method on Zin Deficiency and Dampness Type Polycystic Ovary Syndrome: a Multi-center, Double-blind, Randomized and Placebo-controlled Study
Brief Title: Clinical and Basic Research on the Treatment of Polycystic Ovary Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangxi University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Ruining Liang, chief physician, Jiangxi University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S2018ZPYFE0937
Record Dates: First submitted 2019-09-29; First posted 2019-10-09 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapy group (Experimental)
  Interventions: Drug: Zishen Qingre Lishi Huayu Granules
- Control group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zishen Qingre Lishi Huayu Granules — The treatment group used Zishen Qingre Lishi Huayu Granules, including Zhimu（Anemarrhena asphodeloides Bge.）, Shengdi（Rehmannia glutinosa Libosch.）, Maidong（Ophio pogon japonicus (L.f) KerGawl.） , Bixie（Dioscorea septemloma Thunb.）, Huanglian（Coptis chinensis Franch.）, Zhuling（Polyporus umbellatus（Pers.）Fries）, Xuanshen（Scrophularia ningpoensis Hemsl.）, Zelan（Lycopus lucidus Turcz. Var. Hirtus Regel）, Danshen（Salvia miltiorrhiza Beg.）， Gancao（Glycyrrhiza uralensis Fisch.）. Subjects take the drug from the first day of inclusion. Take 1 pack each time, bid, for 3 months.
  Arms: Therapy group
Drug: Placebo — The treatment group used Caramel pigment、 Ku Ding Cha Extracts、Maltodextrin、Starch and 5% Zishen Qingre Lishi Huayu Granules .
  Subjects take the drug from the first day of inclusion. Take 1 pack each time, bid, for 3 months.
  Arms: Control group

SUMMARY:
Polycystic ovary syndrome is the most common endocrine and metabolic disorder in gynecology. Traditional Chinese medicine has a good clinical effect in the treatment of PCOS. We intend to conduct this trial in strict accordance with the requirements of evidence-based medicine, through a multi-center, randomized, controlled study, using a double-blind, randomized, placebo-controlled study design method to clarify that Zishen Qingre Lishi Huayu Recipe restores spontaneous ovulation in PCOS patients. The overall efficacy of improving the characteristics of Kaohsiung and glucose and lipid metabolism is optimal, and high-level evidence-based evidence is obtained to form a diagnosis and treatment plan for promotion.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as PCOS patients, the diagnostic criteria is: modify the Rotterdam criteria. All subjects must have: no ovulation, combined with polycystic ovarian or / and hyperandrogenism.
2. Age: 20 to 40 years old, no maternity requirements.
3. Willing to be treated according to the treatment plan specified in this study.

Exclusion Criteria:

1. Hyperprolactinemia: In the past year, patients with normal levels can be included.
2. Menopausal FSH levels：FSH > 15 mIU/mL. In the past year, patients with normal levels can be included.
3. Patients with thyroid disease: TSH < 0.2 mIU/mL or >5.5 mIU/mL. In the past year, patients with normal levels can be included.
4. Patients with poorly controlled type 2 diabetes:HbA1c>7.0%, or patients receiving antidiabetic drugs.
5. Patients currently diagnosed with severe anemia (HGB <10 g/dL).
6. Patients with a history of alcohol abuse: Alcohol is defined as drinking 14 times a week or more or binge drinking.
7. Currently suspected Cushing's syndrome patients.
8. Patients suspected of having adrenal or ovarian tumors secreting androgen.
9. In patients with hypertension who are currently untreated or have poor blood pressure control, the interval between two blood pressure measurements is ≥ 60 min, systolic blood pressure ≥ 160 mm Hg or diastolic blood pressure ≥ 100 mm Hg.
10. Patients currently diagnosed with metabolic syndrome
11. Take hormonal drugs, Chinese medicine prescriptions and proprietary Chinese medicines in the last 3 months.
12. There is a history of pregnancy in the last 6 weeks.
13. Abortion or production history in the last 6 weeks.
14. A history of breastfeeding in the last 6 months.
15. Patients with a history of deep vein thrombosis, pulmonary embolism or cerebrovascular disease.
16. Patients with severe primary diseases such as cardiovascular, liver, kidney and hematopoietic system, and mental patients
17. Patients who are expected to discontinue treatment during the trial or who are unable to adhere to treatment for 3 months should be excluded.
18. Reluctant to sign the informed consent form for this study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-09-06 (Actual)

PRIMARY OUTCOMES:
Ovulation rate | The 3rd month
  Ovulation rate of each group during the study period Ovulation rate per group = actual total ovulation frequency / total number of cycles (total number of cycles = number of samples).

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Jiangxi University of Traditional Chinese Medicine, Nanchang, Jiangxi, China